CLINICAL TRIAL: NCT02015871
Title: An Extension Long-Term Safety and Tolerability Trial of Degarelix, Following a 1-year Open-Label, Multi-Centre, Randomised, Parallel-group Trial in Which the Efficacy and Safety of Degarelix One-month Dosing Regimen Was Compared With Goserelin in Chinese Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: An Extension Long-term Safety and Tolerability Trial of Degarelix in Chinese Patients With Prostate Cancer
Acronym: PandaExtension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000006A
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix

SUMMARY:
This trial is an open-label, multi-centre, single arm extension for the 000006 trial in Chinese patients with prostate cancer. Eligible patients will receive monthly (28-day intervals) maintenance doses of 80 mg (20 mg/mL) degarelix administered by subcutaneous (s.c.) injection for a period of 2 years from first visit in this extension trial. Patients, who received goserelin treatment in the main trial, will get a degarelix starting dose (240 mg; 40 mg/mL) at the first visit and continue on degarelix treatment. The purpose of this 2-year extension trial is to collect long-term safety and tolerability data for the one-month dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent before any trial-related activity is performed. A trial-related activity is defined as any procedure that would not have been performed during the normal management of the patient
* Has completed the 000006 trial

Exclusion Criteria:

* Has been withdrawn/discontinued from the 000006 trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with Adverse Events (AEs) | Baseline to Month 26
Change in ECG parameters | Baseline to Month 26
Change in body weight and vital signs | Baseline to Month 26
Clinically significant changes in laboratory values (clinical chemistry, haematology, and urinalysis) | Baseline to Month 26

SECONDARY OUTCOMES:
Change in testosterone levels | Baseline to Month 26
Change in prostate-specific antigen (PSA) levels | Baseline to Month 26
Cumulative probability of no PSA failure | Baseline to Month 26
  PSA failure is defined as two consecutive (at least two weeks apart) increases of 50%, and at least 5 ng/mL, compared to nadir (obtained in either trial 000006 or trial 000006A)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Peking University People's Hospital (there may be multiple sites in this country), Beijing, Beijing Municipality, China